CLINICAL TRIAL: NCT03403465
Title: Intratreatment FDG-PET During Radiation Therapy for Gynecologic and Gastrointestinal Cancers ( Adaptive PET II)
Brief Title: Intratreatment FDG-PET During Radiation Therapy for Gynecologic and Gastrointestinal Cancers
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00089619
Record Dates: First submitted 2018-01-11; First posted 2018-01-18 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Cancer of the Cervix; Vulvar Cancer; Esophageal Cancer; Anal Canal Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms; Vulvar Neoplasms; Esophageal Neoplasms; Anal Canal Carcinoma | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm interventional study (Other): Research FDG-PET scan obtained before radiation therapy; a second research FDG-PET scan is obtained at about 3-5 weeks after treatment has started.
  Interventions: Other: FDG PET scan

INTERVENTIONS:
Other: FDG PET scan — At radiation planning subjects will have a PET-CT. The CT scan - also called computerized tomography or just CT - combines a series of X-ray views taken from many different angles to produce cross-sectional images of the bones and soft tissues inside the body. CT scans in planning radiation therapy are standard of care. A PET is a highly specialized imaging technique that uses short-lived radioactive substances (such as FDG a simple sugar labeled with a radioactive atom) to produce three-dimensional colored images of those substances functioning within the body. These images are called PET scans and the technique is termed PET scanning. PET scanning provides information about the body's chemistry not available through other procedures. Unlike CT or MRI (magnetic resonance imaging), techniques that look at anatomy or body form, PET studies metabolic activity or body function.
  Other Names: PET scan

SUMMARY:
This study expands on protocol (NCT01908504"PET adaptive RT") designed to evaluate the utility of adaptive PET-CT planning for radiation therapy (RT). Radiation therapy is used in many malignant diseases as a curative treatment modality. However, critical normal tissue is often in close approximation to disease, and portions of such tissue must receive high doses of radiation for appropriate treatment.

Positron Emission Tomography (PET) adapted radiation therapy, as defined in the current protocol, may allow for a means of determining the eventual response to therapy, at a time point when adaptation of treatment plan may be possible to improve outcomes. This protocol will build upon the findings the previous protocol (NCT01908504 "PET adaptive RT") that evaluated the utility of intra-treatment PET imaging in multiple types of cancers. The current focus will be more specific to certain types of gastrointestinal and gynecologic cancers treated with RT, identified from the prior study to warrant further research.

DETAILED DESCRIPTION:
Intra-treatment PETs have only recently been studied in small pilot series. In rectal cancer, a prospective trial from MSKCC demonstrated that a PET-CT obtained in the second week of neoadjuvant chemoradiotherapy was able to discriminate sub-optimal responders with a sensitivity of 94% and an accuracy of 78%, though the most useful metric was a novel "visual response score" based on interpreting radiologists scoring rather than more established objective data available from PET, like SUV. A study from China in non-small cell lung cancer found that decreases in SUV and MTV on intra-treatment PET-CTs after 40Gy of chemoradiation therapy were significantly greater in patients responding to treatment by post-treatment RECIST criteria. For head and neck cancers, a Belgian study found that intra-treatment SUVmax at 47Gy was associated with significant differences in overall survival. Therefore, there is emerging evidence that an intra-treatment PET may also be of significant prognostic utility, at an early enough time point to potentially alter treatment accordingly.

All participants will be required to complete two research PET scans in addition to standard of care planning CT's for radiation therapy. For all subjects with cancer of the cervix and vulva an intra-treatment PET-CT will be obtained and used to develop a volume adaptive treatment plan for the remainder of the course. Subjects with esophageal and anal canal cancer will have an adapted plan if the treating radiation oncologist determines an adapted plan is clinically relevant.

ELIGIBILITY:
Inclusion Criteria:

Pathologically (histologically or cytologically) proven diagnosis of cervical, vulvar, esophageal and anal canal cancer

Patients with local or regional nodal disease are eligible

Zubrod Performance Status 0, 1, or 2

Age ≥ 18

Negative serum pregnancy test for women of child bearing potential

Patient must sign study-specific informed consent prior to study entry

Exclusion Criteria:

No gross disease visible on imaging at the start of radiotherapy

Contraindication to PET

Complete response by PET achieved with pre-radiation therapy treatment (surgery or chemotherapy)

Breast feeding

Positive serum pregnancy test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-03-27 (Actual); Primary Completion 2028-04-05 (Estimated); Study Completion 2028-04-05 (Estimated)

PRIMARY OUTCOMES:
The number of subjects with benefit from an intra-treatment PET-CT | 4 years
  This benefit lies in the potential to adapt the treatment plan based on an intratreatment PET-CT. This may also be of significant prognostic utility, at an early enough time point to potentially alter treatment accordingly
Pathologic complete response | 4 years
  Pathologic complete response will be collected from pathology reports for subjects who have surgical resection after radiation therapy.
Locoregional control | Day of intra treatment PET-CT/ approx 2-4 hours
  This study will evaluate the prognostic value of intra-treatment functional imaging on clinical relevant tumor endpoints (i.e. locoregional control, freedom from distant metastases, and overall survival).Comparison of intra-treatment FDG-PET indices will identify two groups of responses: PET responses and PET non-responses, which will correlate with prognosis.
Freedom from distant metastases | 4 years
  Subjects will be evaluated in regular follow up with repeat imaging as per the standard of care, or at the treating investigator's discretion. Frequency of follow up will be determined by the standard practice for the disease site and stage.
Measure overall survival (OS) | 4 years
  Subjects will be evaluated in regular follow up with the investigators according to the standard of care for each disease site
Progression free survival (PFS) | 4 years
  Subjects will be evaluated in regular follow up with repeat imaging as per the standard of care for each disease site

SECONDARY OUTCOMES:
Measure the potential sparing of radiation dose to critical normal tissue | 4 years
  An intra-treatment PET volume adaptive treatment plan may allow for additional sparing of normal tissue by identifying regions of tumor response and corresponding reduction in the target volumes i.e. dosimetric differences in normal tissue will be compared between the initial plan and the adapted plan.

CONTACTS AND LOCATIONS:
Overall Officials: Junzo Chino, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No